CLINICAL TRIAL: NCT06863207
Title: Autonomic Reactivity to Restore a Dysregulated Brain-Gut Axis Via Targeted Therapy
Brief Title: Autonomic Reactivity and Personalized Neurostimulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Katja Karrento, Associate Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO00051003; 1R01DK140255-01 (NIH)
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Functional Gastrointestinal Disorders (FGIDs); Cyclic Vomiting Syndrome; Functional Dyspepsia; Dysautonomia
Keywords: autonomic dysfunction; auricular neurostimulation; gastric motor function; gut-directed hypnotherapy
MeSH Terms: conditions — Gastrointestinal Diseases; Familial cyclic vomiting syndrome; Autonomic Nervous System Diseases; Primary Dysautonomias | interventions — Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- PENFS (percutaneous electrical nerve field stimulation) therapy (Experimental): Personalized PENFS therapy x 6 weeks based on weekly autonomic nervous system assessments
  Interventions: Device: Percutaneous electrical nerve field stimulation
- PENFS (percutaneous electrical nerve field stimulation) therapy + Hypnotherapy (Active Comparator): Personalized PENFS therapy x 6 weeks based on weekly autonomic nervous system assessments + adjuntive hypnotherapy
  Interventions: Device: Percutaneous electrical nerve field stimulation; Behavioral: Hypnotherapy

INTERVENTIONS:
Device: Percutaneous electrical nerve field stimulation — Percutaneously nerve stimulator applied to the external auricle weekly for several consecutive weeks of therapy
Behavioral: Hypnotherapy — Gut-directed hypnotherapy delivered via audio recordings
  Arms: PENFS (percutaneous electrical nerve field stimulation) therapy + Hypnotherapy

SUMMARY:
Disorders of gut-brain interaction (DGBI) affect up to 25% of U.S. children. Patients often suffer from disabling, multisystem comorbidities that suggest a common root (sleep disturbances, fatigue, anxiety, etc). Yet, DGBI are defined and treated based on GI symptom origin (cyclic vomiting, dyspepsia, irritable bowel) rather than underlying pathophysiology. Many patients manifest comorbidities suggesting an underlying autonomic nervous system (ANS) dysregulation (palpitations, dizziness, cognitive dysfunction). Unfortunately, due to common features of anxiety and visceral hyperreactivity and lack of obvious pathology, children with DGBI are frequently diagnosed with psychosomatic or 'benign, functional disorders' and treated with empiric antidepressants despite lack of scientific support and risks of serious side effects. Little is known about the underlying brain-gut mechanisms linking these comorbidities. A lack of targeted treatment options naturally follows the paucity of mechanistic data. A dysregulated ANS response circuit via brainstem nuclei is linked to visceral hypersensitivity. As the team's prior research has shown, ANS regulation can be non-invasively measured via several validated indices of cardiac vagal tone. Using the novel vagal efficiency (VE) metric, the investigators have demonstrated inefficient vagal regulation in cyclic vomiting syndrome and pain-related DGBI and that low VE predicts response to non-invasive, auricular percutaneous electrical nerve field stimulation (PENFS) therapy. PENFS targets brainstem vagal afferent pathways and, along with brain-gut interventions such as hypnotherapy, are the only therapies currently proven effective for pediatric DGBI. Individualizing neurostimulation based on sensory thresholds while assessing dynamic ANS reactivity offers a path towards personalized medicine using the most effective therapies to date. This proposal will test the feasibility of an ANS tracking software in assessing real-time, autonomic regulation and providing individualized neurostimulation in children with nausea/vomiting and ANS imbalance.

DETAILED DESCRIPTION:
The investigators hypothesize that children with cyclic vomiting syndrome (CVS) and chronic nausea/vomiting with concurrent symptoms of autonomic nervous system (ANS) dysregulation have reduced vagal efficiency (VE) that can be captured by the ANS Tracker software and modulated via adjustable percutaneous electrical nerve field stimulation (PENFS). Our overall goals are to: 1) expand knowledge on mechanisms of disorders of gut brain interaction involving VE and gastric function, 2) test a software that allows point of care VE assessment, 3) personalize PENFS parameters with real-time assessments of VE and gastric function, 4) combine and assess efficacy of two proven, effective therapies for DGBI that both modulate CNS.

The specific aims of this study are as follows:

Aim 1: Test the feasibility of real-time autonomic nervous system (ANS) tracking in children with nausea/vomiting and ANS dysregulation The investigators will test feasibility of assessing real-time ANS regulation by the VE metric using a novel ANS tracker software in response to posture shifts during PENFS with 1) standard and 2) personalized stimulation parameters based on sensory thresholds in female children with nausea/vomiting.

Aim 2: Compare efficacy and ANS changes with personalized PENFS +/- adjunctive hypnotherapy The investigators will assess outcomes of 6 weeks of personalized PENFS based on sensory threshold (Aim 1) vs. personalized PENFS with adjunctive hypnotherapy via weekly assessments of VE and symptom response. Baseline VE measurements will be correlated with outcomes to assess ability to predict treatment response.

Aim 3: Investigate dynamic gastric function in response to personalized PENFS The investigators will test real-time gastric function pre and post therapy (Aim 2 interventions) by advanced MRI in a subset of female patients vs. healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* 11 to 18 years of age
* English speaking
* meeting Rome IV diagnostic criteria for cyclic vomiting syndrome or functional dyspepsia and willingness to participate and consent/assent to the study
* All subjects will have a constellation of chronic symptoms indicative of autonomic dysfunction for minimum 3 months: postural dizziness/lightheadedness, syncope, palpitations, fatigue, sleep disturbance, thermoregulatory abnormalities and cognitive impairment with upright position +/- abnormal autonomic testing if performed per standard of care as per American Autonomic Society consensus criteria.

Exclusion Criteria:

* Presence of organic disease that may explain symptoms
* Requirement for parenteral nutrition
* Developmental delays precluding accurate symptom report
* Severe dermatological condition or active infection of external or middle ear
* Implanted electrical device
* Severe mental health disorder not controlled by therapy (schizophrenia, bipolar disease, severe depression, post-traumatic distress disorder) and/or psychotic features which could influence symptom report or ANS measurements and result in adverse reactions to hypnosis therapy

Ages: 11 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01-24 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Profile-37 | From enrollment to end of treatment at 6 weeks
  Validated quality of life instrument assessing physical, emotional, and psychosocial functioning in children across 6 domains (subscales). Scores range from 0 (minimum) to 5 (maximum). A lower score indicates improved quality of life for the Anxiety, Depression, Fatigue and Pain Interference domains/subscales. A higher scores indicates improvement in the Physical Function and Peer Relationships subscales. Scores are converted to a T-score where a score of 50 represents the mean.

SECONDARY OUTCOMES:
2. Patient Assessment of upper GastroIntestinal Symptom Severity Index | From enrollment to the end of treatment at 6 weeks.
  Upper gastrointestinal symptoms including symptoms of gastroparesis will be assessed via this 20-item instrument with scores ranging from 0 (minimum) to 5 (maximum). Higher scores indicate worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Katja Karrento, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to share anonymized, IPD including primary outcome data (PAGI-SYM results) through the publicly accessible Vivli Center for Global Clinical Research Data repository, an NIH supported repository and global data-sharing platform that promotes sharing of individual, participant-level clinical data from clinical trials.
Supporting Information: Study Protocol
Time Frame: Scientific data will be made available no later than the time of an associated publication or the end of the performance period (June 2029), whichever comes first. The investigators anticipate that data will be available for approximately 7-10 years, provided that software upgrades during that time allow compatibility.
Access Criteria: Any researcher can access de-identified IPD including study protocol, manual of operations, any data collection forms and results of primary outcome via Vivli Center for Global Clinical Research Data Repository.
URL: https://vivli.org/members/why-we-support-vivli/

REFERENCES:
- [Background] Kolacz J, Roath OK, Lewis GF, Karrento K. Cardiac Vagal Efficiency Is Enhanced by Percutaneous Auricular Neurostimulation in Adolescents With Nausea: Moderation by Antidepressant Drug Exposure. Neurogastroenterol Motil. 2025 May;37(5):e15007. doi: 10.1111/nmo.15007. Epub 2025 Jan 30. PMID 39888101
- [Background] Sclocco R, Garcia RG, Kettner NW, Isenburg K, Fisher HP, Hubbard CS, Ay I, Polimeni JR, Goldstein J, Makris N, Toschi N, Barbieri R, Napadow V. The influence of respiration on brainstem and cardiovagal response to auricular vagus nerve stimulation: A multimodal ultrahigh-field (7T) fMRI study. Brain Stimul. 2019 Jul-Aug;12(4):911-921. doi: 10.1016/j.brs.2019.02.003. Epub 2019 Feb 10. PMID 30803865
- [Background] Kovacic K, Hainsworth K, Sood M, Chelimsky G, Unteutsch R, Nugent M, Simpson P, Miranda A. Neurostimulation for abdominal pain-related functional gastrointestinal disorders in adolescents: a randomised, double-blind, sham-controlled trial. Lancet Gastroenterol Hepatol. 2017 Oct;2(10):727-737. doi: 10.1016/S2468-1253(17)30253-4. Epub 2017 Aug 18. PMID 28826627
- [Background] Menys A, Keszthelyi D, Fitzke H, Fikree A, Atkinson D, Aziz Q, Taylor SA. A magnetic resonance imaging study of gastric motor function in patients with dyspepsia associated with Ehlers-Danlos Syndrome-Hypermobility Type: A feasibility study. Neurogastroenterol Motil. 2017 Sep;29(9). doi: 10.1111/nmo.13090. Epub 2017 May 31. PMID 28568908
- [Background] Holtmann G, Goebell H, Jockenhoevel F, Talley NJ. Altered vagal and intestinal mechanosensory function in chronic unexplained dyspepsia. Gut. 1998 Apr;42(4):501-6. doi: 10.1136/gut.42.4.501. PMID 9616311
- [Background] Lewis GF, Furman SA, McCool MF, Porges SW. Statistical strategies to quantify respiratory sinus arrhythmia: are commonly used metrics equivalent? Biol Psychol. 2012 Feb;89(2):349-64. doi: 10.1016/j.biopsycho.2011.11.009. Epub 2011 Dec 3. PMID 22138367
- [Background] Kovacic K, Kolacz J, Lewis GF, Porges SW. Impaired Vagal Efficiency Predicts Auricular Neurostimulation Response in Adolescent Functional Abdominal Pain Disorders. Am J Gastroenterol. 2020 Sep;115(9):1534-1538. doi: 10.14309/ajg.0000000000000753. PMID 32732620
- [Background] Kolacz J, Kovacic K, Dang L, Li BUK, Lewis GF, Porges SW. Cardiac Vagal Regulation Is Impeded in Children With Cyclic Vomiting Syndrome. Am J Gastroenterol. 2023 Jul 1;118(7):1268-1275. doi: 10.14309/ajg.0000000000002207. Epub 2023 Jan 30. PMID 36716443
- [Background] Venkatesan T, Prieto T, Barboi A, Li B, Schroeder A, Hogan W, Ananthakrishnan A, Jaradeh S. Autonomic nerve function in adults with cyclic vomiting syndrome: a prospective study. Neurogastroenterol Motil. 2010 Dec;22(12):1303-7, e339. doi: 10.1111/j.1365-2982.2010.01577.x. PMID 20667005
- See also: Global clinical research data sharing platform that will be used as repository to share participant-level data once results are available. — https://vivli.org/
- Available data/document: Individual Participant Data Set — https://vivli.org/